CLINICAL TRIAL: NCT05859906
Title: Evaluation of the Effect of Two Different Intra-abdominal Pressure Applications on "Mechanical Power" in Cases Undergoing Laparoscopic Cholecystectomy
Brief Title: The Effect of Two Different Intra-abdominal Pressure Applications on "Mechanical Power" in Laparoscopic Cholecystectomy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ayse Ulgey (Other)
Responsible Party: Sponsor-Investigator, Ayse Ulgey, Professor Doctor, TC Erciyes University
Organization: TC Erciyes University (Other)
Other Study IDs: 2023/104
Record Dates: First submitted 2023-05-05; First posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Ventilator-induced Lung Injury
Keywords: Mechanical power; laparoscopic surgery; Ventilator-induced lung injury
MeSH Terms: conditions — Ventilator-Induced Lung Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 12 mmHg: All patients in this group will be operated with an insufflation pressure of 12 mmHg during laparoscopic cholecystectomy surgery.
  Interventions: Other: mechanical power measurement
- Group 14 mmHg: All patients in this group will be operated with an insufflation pressure of 14 mmHg during laparoscopic cholecystectomy surgery.
  Interventions: Other: mechanical power measurement

INTERVENTIONS:
Other: mechanical power measurement — Mechanical power values of the patients;
  * Before insufflation (baseline value),
  * 0 min after insufflation,
  * 15th min after insufflation,
  * 30 minutes after insufflation,
  * 45th minute after insufflation (if insufflation continues),
  * 60th minute after insufflation (if insufflation continues),
  * Intraoperative after insufflation It will be measured with the following formula in the specified periods. MP = 0.098 x minute ventilation x [Peak inspiratory pressure - 0.5 x (Plateau pressure - Positive end-expiratory pressure)]

SUMMARY:
In laparoscopic surgeries; a trocar is inserted through a small incision and an intervention is made into the peritoneal cavity. Approximately 3-4 liters of carbon dioxide (CO2) insufflation (inflating the abdominal cavity with carbon dioxide gas) is applied and the intra-abdominal pressure is adjusted to 10-20 mmHg. Laparoscopic cholecystectomy operation is routinely performed with 12 mmHg and 14 mmHg pressures in our operating room, and the preferred pressure value is; It is determined by the surgical team to be the most appropriate value for the patient and the operation. Both pressure values applied to the patients intraoperatively are within safe ranges.

The mechanical power of ventilation (MP) is the amount of energy transferred per unit time from the mechanical ventilator to the respiratory system. Although this energy is mainly used to overcome airway resistance, some of it directly affects the lung tissue, potentially causing ventilator induced lung injury (VILI). To prevent ventilator-associated lung injury, it requires the mechanical ventilator to be adjusted so that the least amount of energy is transferred to the respiratory system per unit time for each patient. In the results obtained in the published studies; increased mechanical strength has been associated with increased in-hospital mortality, higher hospital stay and higher ICU follow-up requirement.

The aim of this study is to investigate the effect of two different intra-operative intra-abdominal pressure levels applied to patients who underwent laparoscopic cholecystectomy under general anesthesia on 'Mechanical Power (MP)'.

DETAILED DESCRIPTION:
In laparoscopic surgeries; a trocar is inserted through a small incision and an intervention is made into the peritoneal cavity. Approximately 3-4 liters of carbon dioxide (CO2) insufflation (inflating the abdominal cavity with carbon dioxide gas) is applied and the intra-abdominal pressure is adjusted to 10-20 mmHg. Intra-abdominal pressure is continuously measured by pressure monitoring, which is routinely performed during laparoscopic procedures. The applied intra-abdominal pressure is determined by the surgical team and the most optimal value that creates pneumoperitoneum for the patient is preferred. Abdominal compartment syndrome can be seen due to abdominal hypertension at intra-abdominal pressure values above 20 mmHg.

Both pressure values aimed to be applied in this study are applied in laparoscopic cholecystectomy operations and do not cause any harm to the patient and their superiority to each other has not been determined.

Laparoscopic cholecystectomy operation is routinely performed with 12 mmHg or 14 mmHg pressures in our operating room. Both pressure values applied to the patients intraoperatively are within safe ranges.

The mechanical power of ventilation (MP) is the amount of energy transferred per unit time from the mechanical ventilator to the respiratory system. Although this energy is mainly used to overcome airway resistance and respiratory system compliance, some of it directly affects the lung tissue, potentially causing ventilator induced lung injury (VILI).

MP is a summary variable that includes several components, including tidal volume (VT ), peak pressure (Ppeak), driving pressure (Driving Pressure, ΔP), and respiratory rate (RR). These components; requires that the mechanical ventilator be adjusted so that the least amount of energy is transferred to the respiratory system per unit time for each patient in order to prevent ventilator-associated lung injury.

In the researches; a relationship between mechanical power (MP) and complications such as ventilator-associated lung injury (VILI) and acute respiratory distress syndrome (ARDS) has been found. The findings suggest that the mechanical force applied to the lungs should be reduced during intraoperative ventilation in patients undergoing major surgery. In adult patients undergoing general anesthesia during major surgical operations, higher patient exposure to ventilation as measured by higher mechanical power; it has been shown that it is associated with an increased risk of postoperative pulmonary complications and acute respiratory failure in the first 7 days of the postoperative period.

In the results obtained in the published studies; increased mechanical strength has been associated with increased in-hospital mortality and higher hospital stay and higher ICU follow-up requirement.

The aim of this study is to investigate the effect of two different intra-operative intra-abdominal pressure levels applied to patients who underwent laparoscopic cholecystectomy under general anesthesia on 'Mechanical Power (MP)'.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ASA 1-2
* The patient's willingness to participate in the study voluntarily

Exclusion Criteria:

* Patients with ASA 3-4
* Patients with lung disease such as pneumonia, COPD attack before the operation
* Patients undergoing other surgical procedures or anesthesia technique
* Pregnant patients
* Patients with morbid obesity
* Unstable patients such as uncontrolled hypertension, decompensated heart disease
* The patient's intraoperative intra-abdominal pressure value is operated with a difference from the pressure determined due to optimal surgical conditions or the patient's lungs do not tolerate it, or switching to open surgery (laparotomy) for any reason.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 200 patients who will be operated for laparoscopic cholecystectomy at Erciyes University between May 2023 and Oct 2023 will be included in our study.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-05-15 (Estimated); Primary Completion 2023-08-15 (Estimated); Study Completion 2023-10-15 (Estimated)

PRIMARY OUTCOMES:
ventilator-induced lung injury (barotrauma) | during the operation
  mechanical power values measured during operation will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Ülgey, MD, Study Director — TC Erciyes University
Locations (1):
- Ayşe Ülgey, Kayseri, Talas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identifed individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 6 months of study completion
Access Criteria: Data accept requests will be reviewed by an external independent Review Panel. Requesters will be required to sign a Data Access Agreement

REFERENCES:
- [Background] Protti A, Andreis DT, Monti M, Santini A, Sparacino CC, Langer T, Votta E, Gatti S, Lombardi L, Leopardi O, Masson S, Cressoni M, Gattinoni L. Lung stress and strain during mechanical ventilation: any difference between statics and dynamics? Crit Care Med. 2013 Apr;41(4):1046-55. doi: 10.1097/CCM.0b013e31827417a6. PMID 23385096
- [Background] Cressoni M, Gotti M, Chiurazzi C, Massari D, Algieri I, Amini M, Cammaroto A, Brioni M, Montaruli C, Nikolla K, Guanziroli M, Dondossola D, Gatti S, Valerio V, Vergani GL, Pugni P, Cadringher P, Gagliano N, Gattinoni L. Mechanical Power and Development of Ventilator-induced Lung Injury. Anesthesiology. 2016 May;124(5):1100-8. doi: 10.1097/ALN.0000000000001056. PMID 26872367
- [Background] Gattinoni L, Tonetti T, Cressoni M, Cadringher P, Herrmann P, Moerer O, Protti A, Gotti M, Chiurazzi C, Carlesso E, Chiumello D, Quintel M. Ventilator-related causes of lung injury: the mechanical power. Intensive Care Med. 2016 Oct;42(10):1567-1575. doi: 10.1007/s00134-016-4505-2. Epub 2016 Sep 12. PMID 27620287
- [Background] Karalapillai D, Weinberg L, Neto A S, Peyton P, Ellard L, Hu R, Pearce B, Tan CO, Story D, O'Donnell M, Hamilton P, Oughton C, Galtieri J, Wilson A, Eastwood G, Bellomo R, Jones DA. Intra-operative ventilator mechanical power as a predictor of postoperative pulmonary complications in surgical patients: A secondary analysis of a randomised clinical trial. Eur J Anaesthesiol. 2022 Jan 1;39(1):67-74. doi: 10.1097/EJA.0000000000001601. PMID 34560687
- Available data/document: Clinical Study Report — http://doi.org/10.1093/bjaceaccp/mkh037